CLINICAL TRIAL: NCT02876965
Title: Change on Sleep Quality of Patients With Fibromyalgia Subjected to a Combined Protocol Based on Physical Exercise and Muscle Stretching
Brief Title: Change on Sleep Quality of Patients With Fibromyalgia Subjected to a Protocol Based on Physical Exercise and Stretching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Fco. Javier Montanez Aguilera, PhD, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU-UCH
Record Dates: First submitted 2016-08-14; First posted 2016-08-24 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Fibromyalgia; Sleep; Stretch
MeSH Terms: conditions — Fibromyalgia | interventions — Muscle Stretching Exercises; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Exercise (Active Comparator): Aerobic physical exercise protocol of moderate intensity, for 12 weeks, 3 sessions per week, about 12 minutes. Physical activity chosen will be pedaling on a static bike.
  Interventions: Procedure: Physical Exercise
- Muscle Stretching (Experimental): Stretching program on the main muscle groups of the body, for 12 weeks, 1sessions per week, about 45 minutes.
  Interventions: Procedure: Muscle Stretching; Procedure: Physical Exercise

INTERVENTIONS:
Procedure: Muscle Stretching — Subjects completed one stretching session on the main muscle groups of the body weekly.
  Arms: Muscle Stretching
Procedure: Physical Exercise — Subjects completed 3 moderate intensity aerobic physical exercise sessions weekly.

SUMMARY:
This study evaluates the effect to a muscle stretching program combined with physical exercise versus a physical exercise program in patients with fibromyalgia.

DETAILED DESCRIPTION:
Although classically this pathology was characterized by having an unknown etiology, current research suggests that the disease shows several abnormalities in the central pain processing.

Central sensitization is defined as changes in neuroplasticity of central nervous system as a result of persistent and intense sensory information nociceptive generated by peripheral and transmitted to the neurons in the dorsal horn of the cord through the nerves of the peripheral nervous system tissues, through a constant activity of C fibers and A-beta fibers.

In recent years the theory that pain is responsible for other symptoms, is changing, and it is theorized that the quality of sleep directly influences in the symptoms.

The treatment of fibromyalgia is based on trying to reduce pain and associated symptoms described above in order to improve the quality of life of these patients. Almost all revisions studying the effects of physical activity in fibromyalgia agree that it is effective in reducing the overall impact on the disease and its symptoms.

Muscle strength training aim to improve the strength, endurance and muscle power. There are few conclusive studies on the benefits of stretching and flexibility exercises on the impact of fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or more.
* To be diagnosed with fibromyalgia according to the criteria established by the "American College of Rheumatology", either on the basis of its publication of 1990 or the current revision of 2010.
* Accept to volunteer and give oral consent. Before starting the intervention must be provided written informed consent.

Exclusion Criteria:

* Do not present any pathology in which physical exercise is contraindicated.
* Do not suffer another serious somatic illness or severe psychological disorder. Not suffer severe dementia (MMSE <10).
* Do not be participating at the time of the study in any other intervention of physical or psychological.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index | At the beginning, every two weeks up to 12 weeks
  The Pittsburgh Sleep Quality Index, where a lower score (0-21), better sleep quality. Follows a continuous metric scale.

SECONDARY OUTCOMES:
Epworth sleepiness scale | At the beginning, every two weeks up to 12 weeks
  The Epworth Sleepiness Scale, where a lower score (0-24), better sleep. Follows a continuous metric scale.
Sleep scale (medical outcomes study) | At the beginning, every two weeks up to 12 weeks
  The Sleep Scale from the Medical Outcomes Study evaluates the quality of sleep with a score of (0-100), where 0 is "no problem" and 100 is "maximum problems". Follows a continuous metric scale.
Visual analog scale | At the beginning, every two weeks up to 12 weeks
  The visual analog scale measures the perceived pain with a score ofh a (0-100), where a higher score means more pain. Follows a continuous metric scale.
Fibromyalgia impact questionnaire | At the beginning, every two weeks up to 12 weeks
  The Fibromyalgia Impact Questionnaire follows a continuous metric scale, (0-100), where a higher score means lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: F Javier Montañez-Aguilera, PhD, Principal Investigator — CEU Cardenal Herrera University
Locations (1):
- CEU Cardenal Herrera University, Moncada, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Result] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Result] Clauw DJ. Fibromyalgia: an overview. Am J Med. 2009 Dec;122(12 Suppl):S3-S13. doi: 10.1016/j.amjmed.2009.09.006. PMID 19962494
- [Result] Gormsen L, Rosenberg R, Bach FW, Jensen TS. Depression, anxiety, health-related quality of life and pain in patients with chronic fibromyalgia and neuropathic pain. Eur J Pain. 2010 Feb;14(2):127.e1-8. doi: 10.1016/j.ejpain.2009.03.010. Epub 2009 May 26. PMID 19473857
- [Result] Shah MA, Feinberg S, Krishnan E. Sleep-disordered breathing among women with fibromyalgia syndrome. J Clin Rheumatol. 2006 Dec;12(6):277-81. doi: 10.1097/01.rhu.0000249771.97221.36. PMID 17149057
- [Result] Moldofsky H. Rheumatic manifestations of sleep disorders. Curr Opin Rheumatol. 2010 Jan;22(1):59-63. doi: 10.1097/BOR.0b013e328333b9cc. PMID 19935069
- [Result] Moldofsky H. The significance, assessment, and management of nonrestorative sleep in fibromyalgia syndrome. CNS Spectr. 2008 Mar;13(3 Suppl 5):22-6. doi: 10.1017/s1092852900026808. PMID 18323770
- [Result] Valkeinen H, Hakkinen A, Hannonen P, Hakkinen K, Alen M. Acute heavy-resistance exercise-induced pain and neuromuscular fatigue in elderly women with fibromyalgia and in healthy controls: effects of strength training. Arthritis Rheum. 2006 Apr;54(4):1334-9. doi: 10.1002/art.21751. PMID 16575859
- [Result] Jones KD, Adams D, Winters-Stone K, Burckhardt CS. A comprehensive review of 46 exercise treatment studies in fibromyalgia (1988-2005). Health Qual Life Outcomes. 2006 Sep 25;4:67. doi: 10.1186/1477-7525-4-67. PMID 16999856
- [Result] Busch AJ, Barber KA, Overend TJ, Peloso PM, Schachter CL. Exercise for treating fibromyalgia syndrome. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD003786. doi: 10.1002/14651858.CD003786.pub2. PMID 17943797